CLINICAL TRIAL: NCT05788094
Title: Does Artemisinin Combination Treatment Reduce the Radical Curative Efficacy of High Dose Tafenoquine for Plasmodium Vivax Malaria?
Brief Title: ACT vs CQ With Tafenoquine for P. Vivax Mono-infection
Acronym: ACTQ
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shoklo Malaria Research Unit (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, SMRU, Dr Aung Pyae Phyo, Associate Research Fellow, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMRU-01/23
Record Dates: First submitted 2023-01-09; First posted 2023-03-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Malaria; Malaria, Vivax; Plasmodium Vivax Malaria
Keywords: artemisinin combination treatment; tafenoquine; Plasmodium vivax malaria; Malaria
MeSH Terms: conditions — Malaria; Malaria, Vivax | interventions — tafenoquine; Chloroquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: Randomised open label non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dihydroartemisinin-piperaquine plus tafenoquine (450 mg adult dose) (Experimental): * Dihydroartemisinin-Piperaquine will be purchased as Duo-Cotecxin® Beijing Holley-Cotec Pharmaceuticals Co., Ltd, China). One tablet contains 40 mg of dihydroartemisinin and 320 mg piperaquine (i.e. a 1:8 ratio). A weight-based regimen containing a total dose of approximately 7 mg/kg DHA and 55 mg/kg piperaquine given in 3 divided doses once daily.
  * Tafenoquine KODATEF® 100 mg film-coated tablets will be purchased from Biocelect (Suite 5.02, Level 5, 139 Macquarie Street, Sydney NSW, 2000 Australia), 450 mg (4 1/2 tablets) will be given.
  Interventions: Drug: Dihydroartemisinin-piperaquine plus tafenoquine (450 mg adult dose)
- Chloroquine plus Tafenoquine (450 mg adult dose) (Experimental): * Chloroquine will be dosed as a 25 mg/kg base given in divided doses of 10 mg/kg orally on days 0 and 1, and in 5 mg/kg dose on day 2. Tablets will be obtained from Government Pharmaceutical Organization (GPO) in Bangkok, Thailand and supplied as 250 mg tablets (155.3 mg base).
  * Tafenoquine KODATEF® 100 mg film-coated tablets will be purchased from Biocelect (Suite 5.02, Level 5, 139 Macquarie Street, Sydney NSW, 2000 Australia), 450 mg (4 1/2 tablets) will be given.
  Interventions: Drug: Chloroquine plus Tafenoquine (450 mg adult dose)
- Artemether-Lumefantrine plus Tafenoquine (450 mg adult dose) (Experimental): * Artemether-Lumefantrine will be given at a standard dose of 20/120 mg twice daily for three days. (AL will be purchase from Novartis Pharma Services AG- Lichtstrasse 35, CH-4056 Basel, Switzerland.)
  * Tafenoquine KODATEF® 100 mg film-coated tablets will be purchased from Biocelect (Suite 5.02, Level 5, 139 Macquarie Street, Sydney NSW, 2000 Australia), 450 mg (4 1/2 tablets) will be given.
  Interventions: Drug: Artemether-Lumefantrine plus Tafenoquine (450 mg adult dose)

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine plus tafenoquine (450 mg adult dose) — * Dihydroartemisinin-Piperaquine will be purchased as Duo-Cotecxin® Beijing Holley-Cotec Pharmaceuticals Co., Ltd, China). One tablet contains 40 mg of dihydroartemisinin and 320 mg piperaquine (i.e. a 1:8 ratio). A weight-based regimen containing a total dose of approximately 7 mg/kg DHA and 55 mg/kg piperaquine given in 3 divided doses once daily.
  * Tafenoquine KODATEF® 150 mg film-coated tablets will be purchased from Biocelect (Suite 5.02, Level 5, 139 Macquarie Street, Sydney NSW, 2000 Australia), 450 mg (4 1/2 tablets) will be given.
  Arms: Dihydroartemisinin-piperaquine plus tafenoquine (450 mg adult dose)
Drug: Chloroquine plus Tafenoquine (450 mg adult dose) — * Chloroquine will be dosed as a 25 mg/kg base given in divided doses of 10 mg/kg orally on days 0 and 1, and in 5 mg/kg dose on day 2. Tablets will be obtained from Government Pharmaceutical Organization (GPO) in Bangkok, Thailand and supplied as 250 mg tablets (155.3 mg base).
  * Tafenoquine KODATEF® 150 mg film-coated tablets will be purchased from Biocelect (Suite 5.02, Level 5, 139 Macquarie Street, Sydney NSW, 2000 Australia), 450 mg (4 1/2 tablets) will be given.
  Arms: Chloroquine plus Tafenoquine (450 mg adult dose)
Drug: Artemether-Lumefantrine plus Tafenoquine (450 mg adult dose) — * Artemether-Lumefantrine will be given at a standard dose of 20/120 mg twice daily for three days. (AL will be purchase from Novartis Pharma Services AG- Lichtstrasse 35, CH-4056 Basel, Switzerland.)
  * Tafenoquine KODATEF® 100 mg film-coated tablets will be purchased from Biocelect (Suite 5.02, Level 5, 139 Macquarie Street, Sydney NSW, 2000 Australia), 450 mg (4 1/2 tablets) will be given.
  Arms: Artemether-Lumefantrine plus Tafenoquine (450 mg adult dose)

SUMMARY:
In this area of Greater Mekong Subregion (GMS), vivax malaria is the most common kind of malaria. It can stay very long in the liver, and come out later to make another episode of illness. This can happen many times even without a mosquito bite. Only 8-aminoquinoline drugs can kill the liver forms of the malaria parasite. One of these drugs is called primaquine, and it has been used all over the world for a long time. There is now a new formulation of this 8-aminoquinoline drug called tafenoquine that can also treat the malaria in the liver. The main benefit of this drug is that it is a single dose, which makes much convenient for the patients as well as for the malaria control program than conventional 14 days of primaquine. Recent research suggests that ACT (Artemisinin Combination Therapy) may antagonise the efficacy of tafenoquine (Baird et al. 2020 ASTMH Annual Meeting) . This could prevent the use of tafenoquine in areas with chloroquine resistant P. vivax parasites where national malaria programmes recommend ACTs for vivax malaria. Also, currently recommended tafenoquine dose is sub-optimal: 300 mg dose proved significantly inferior to low dose primaquine in a meta-analysis of the phase 3 studies when restricted to the Southeast Asian region (Llanos-Cuentas et al. 2019 NEJM; Watson et al. 2022a Elife). A tafenoquine dose of 450mg is predicted to provide >90% of the maximal effect. The objective of this research is to find out whether 450 mg dose of tafenoquine can be combined effectively with ACT providing a short course treatment for P. vivax malaria.

DETAILED DESCRIPTION:
Plasmodium vivax malaria is a major cause of morbidity and is a significant contributor to mortality in tropical regions (Battle et al. 2019 The Lancet). Relapses are the major cause of illness and in higher transmission settings contribute to severe anaemia and death in young children as well as pregnancy loss.

SE Asia has the highest proportion of the estimated global burden of P. vivax malaria burden 51.2% (7.2 million of 14.3 million) in 2017.

In SE Asia over half of the patients treated for an acute P. vivax blood stage infection will develop at least one relapse (Betuela et al. 2012 J. Infect. Dis.; Chu et al. 2018 Clin. Infect. Dis.; Commons et al. 2019 BMC Med; Luxemburger et al. 1999 Trans R Soc Trop Med Hyg; Poespoprodjo et al. 2009 Clin. Infect. Dis.; Sutanto et al. 2013 AAC) if an anti-relapse drug is not given. The only widely available drug to prevent relapses (radical cure) currently is the 8-aminoquinoline primaquine. The doses of primaquine required to prevent relapses in Southeast Asia and the Western Pacific region are higher than elsewhere. P. vivax relapses more in these regions where with large populations over 80% of the global P. vivax burden occurs so it is likely that most of the world's relapses occur in East Asia and thus the benefits of effective radical cure are greatest in this area.

Adherence to the currently recommended 14-day primaquine regimen is variable and this compromises widespread primaquine use and efficacy (Cheoymang et al. 2015 Acta tropica; Grietens et al. 2010 ASTMH; Leslie et al. 2004 Trans R Soc Trop Med Hyg; Maneeboonyang et al. 2011 Southeast Asian J. Trop. Med. Public Health) . Recently a slowly eliminated 8-aminoquinoline, tafenoquine, has become available and has been registered in several countries. Tafenoquine can be given in a single dose (Lacerda et al. 2019 NEJM; Llanos-Cuentas et al. 2014a The Lancet; Llanos-Cuentas et al. 2019 NEJM) which allows supervised dosing. However, tafenoquine is contraindicated in persons with G6PD activity below 70% as it may cause significant haemolysis in G6PD deficiency (including in female heterozygotes who may test as normal with current qualitative screens). Thus, quantitative G6PD deficiency testing is required to identify individuals with intermediate G6PD activity to ensure that female G6PD deficiency heterozygotes are not enrolled. Near patient quantitative G6PD tests (G6PD Biosensor) (Bancone et al. 2018 PLoS One; Pal et al. 2019 ASTMH; Zobrist et al. 2021 PLOS Negl. Trop. Dis.) which provide a quantitative result will be used before tafenoquine is prescribed.

The currently recommended tafenoquine dose is sub-optimal. The 300 mg dose proved significantly inferior to low dose primaquine in a meta-analysis of the phase 3 studies when restricted to the Southeast Asian region (Llanos-Cuentas et al. 2019 NEJM; Watson et al. 2022a Elife).

These data and an individual patient data meta-analysis of all (>1000) patients in the pre-registration studies (J. A.Watson et al. 2022a Elife) suggest that a 450mg adult dose of tafenoquine is needed in the Southeast Asian and Western Pacific regions. Doses up to 1200mg have proved safe and well tolerated in G6PD normal individuals.

However a recent study suggests that ACTs may antagonize the curative efficacy of tafenoquine. If true this would complicate current treatment of both falciparum and vivax malaria with a single blood stage drug. The results from the INSPECTOR trial in Indonesian soldiers returning to non-endemic areas showed very low radical curative efficacy with tafenoquine in combination with DHA-PPQ (21%) - an efficacy which was similar to DHA-PPQ alone (11%) (Baird et al. 2020 ASTMH Annual meeting).

This has prompted a product label update for Krintafel® (the branded form of tafenoquine in the USA) that tafenoquine should be combined only with chloroquine and not with other antimalarials such as artemisinin-based combination therapies (ACT)(CDC 2020). This now prevents the use of tafenoquine in areas with chloroquine resistant P. vivax parasites where national malaria programmes recommend ACTs for vivax malaria. As chloroquine resistance in P. vivax is increasing this poses a serious challenge to the potential use of this new radical cure antimalarial. However, this result is at variance with our earlier studies with the structurally and mechanistically similar primaquine, where radical curative efficacies were similar with ACTs (either DHA-PPQ or AL) and chloroquine combinations (Chu et al. 2019 Clin. Infect. Dis.). Whether DHA-PPQ or AL can be combined effectively with tafenoquine needs to be resolved quickly to guide deployment.

Tafenoquine could be particularly valuable in conflict-torn Myanmar where vivax malaria is now out of control and health services have broken down. This clinical trial will be performed in the clinics and health centres in Myawaddy district supervised by Shoklo Malaria Research Unit.

Scientific Rationale

Tafenoquine, as a single dose regimen, has a tremendous advantage over the longer courses of primaquine needed for radical cure. Its use will be progressively restricted if it cannot be used in combination with ACTs. This trial will assess whether or not ACTs (either AL or DHA-PPQ) significantly reduces tafenoquine radical curative efficacy in comparison with chloroquine.

Data Sharing

Paper records will be preserved for five years. Electronic data will be de-identified and preserved indefinitely. With participant's consent, clinical data and results from blood analyses stored in the database may be shared according to the terms defined in the data sharing policy (available at: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing) with other researchers to use in the future.

All personal information will be anonymised so that no individual can be identified from their treatment records. The genomic data sharing plan will be shared on a public database and the plan will be kept in the Regulatory Binder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with P. vivax mono-infection as diagnosed by Rapid Diagnostic Test
* Fever or history of fever in the previous 7 days
* Quantitative G6PD activity ≥70% of the population median i.e., ≥6.1U/gHb
* Age > 18 years, Weight >35 kg
* Ability to understand the study instructions and provide informed consent
* Willing to be followed for 4 months and likely to adhere to the study protocol.

Exclusion Criteria:

* Coincident P. falciparum malaria or other infections
* Pregnancy
* Lactation
* Hb < 8 g/dL
* Quantitative G6PD activity <70% of the population median i.e., <6.1U/gHb
* Severe malaria (as per WHO guideline)
* History of allergic or haemolytic response to any of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Determine whether ACTs (Artemether-Lumefantrine or dihydroartemisinin-piperaquine (DHA-PPQ)) plus TQ is non-inferior to CQ plus TQ | Month-4
  Number of participants with relapse-free efficacy (measured by PCR) in three arms

SECONDARY OUTCOMES:
Characterise the safety and tolerability of three regimens | Day3, Day7, Month1, Month2, Month3, Month4
  Number of participants with drop in hemoglobin ≥2 g/dL and/or hematocrit by ≥10% from baseline
  Number of participants with Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Characterise population pharmacokinetics of tafenoquine in three treatments | Day3, Day7, Month1, Month2, Month3, Month4
  Area Under the Curve From Time-0 Extrapolated to Infinite Time (AUC0-infinite time) of Tafenoquine
Met-Haemoglobin level a vivo pharmacodynamic proxy of oxidative antimalarial activity of tafenoquine | Day3, Day7
  Percentage increase in Methaemoglobin level compared across three arms

OTHER OUTCOMES:
Genotyping and probabilistic assessment to differentiate P. vivax relapse from reinfection | Day3, Day7, Month1, Month2, Month3, Month4
  Number of participants with relapse and reinfection in three regimens
Evaluate the performance of village health workers as safe prescribers of tafenoquine radical cure | Day3, Day7, Month1, Month2, Month3, Month4
  Number of participants with correct dosing, adverse event recording including haemoglobin drops

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, Prof, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Mae Sot, Changwat Tak, Thailand